CLINICAL TRIAL: NCT06806930
Title: Predicting Response to Neoadjuvant Endocrine Therapy (Neo-PREDICT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Pavani Chalasani, Professor of Medicine; Director, Division of Hematology Oncology, George Washington University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neo-PREDICT
Record Dates: First submitted 2025-01-15; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Carcinoma, Breast
Keywords: breast; cancer; HER2; carcinoma
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Carcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A: Short Duration NET (Active Comparator): Patients in this cohort can be treated with NET up to 8weeks (<= 8 weeks)
  Interventions: Drug: Neoadjuvant endocrine therapy
- Cohort B: Intermediate Duration NET (Active Comparator): Patients in this cohort can be treated with NET > 8weeks but <=24 weeks
  Interventions: Drug: Neoadjuvant endocrine therapy
- Cohort C: Extended Duration NET (Active Comparator): Patients in this cohort can be treated with NET >24 weeks but <= 52 weeks
  Interventions: Drug: Neoadjuvant endocrine therapy

INTERVENTIONS:
Drug: Neoadjuvant endocrine therapy — Cohort A: Short duration NET. Patients in this cohort can be treated with NET up to 8weeks (<= 8 weeks)
  Arms: Cohort A: Short Duration NET
Drug: Neoadjuvant endocrine therapy — Cohort B: Intermediate duration NET. Patients in this cohort can be treated with NET > 8weeks but <=24 weeks
  Arms: Cohort B: Intermediate Duration NET
Drug: Neoadjuvant endocrine therapy — Cohort C: Extended duration NET. Patients in this cohort can be treated with NET >24 weeks but <= 52 weeks
  Arms: Cohort C: Extended Duration NET

SUMMARY:
The goal of this clinical trial is to determine how the duration of hormone blocking (endocrine) therapy given prior to surgery (called "neoadjuvant" treatment) affects breast cancer. The main questions the trial aims is answer are:

1. How breast cancer responds to endocrine therapy given prior to surgery?
2. To predict tumor pre-operative endocrine prognostic index (PEPI) score for subjects enrolled in cohort B or C

Participants with early-stage breast cancer (Stage I-III) who are eligible for Neoadjuvant Endocrine Therapy (NET) will be enrolled in the study. Participants will:

* receive endocrine therapy as part of regular care for breast cancer
* consent to samples of blood and tissue evaluation to determine how endocrine therapy effects the tumor
* participate in this research anywhere from 2 weeks to 1 year, depending on duration of endocrine therapy and when surgery will be performed

ELIGIBILITY:
Inclusion Criteria:

* Be capable of understanding the investigational nature of the study and all pertinent aspects of the study
* Be capable of signing and providing written consent in accordance with institutional and federal guidelines
* Histologically or cytologically confirmed diagnosis of invasive carcinoma of the breast
* Clinical stage 1 to 3 breast cancer
* Candidate for surgical resection
* Estrogen receptor > 10% positive stained cells based on most recent tumor biopsy and documented by a local laboratory or medical record.
* HER2 negative or HER2 low breast cancer based on the most recent tumor biopsy and documented by a local laboratory or medical record. HER2 negative tumor is defined per American Society of Clinical Oncology and the College of American Pathologists guidelines, 2018. Patients with HER2 low tumors are eligible as long as patients are not candidates for any HER2 directed therapy.
* Ability to take oral medication
* Be willing and able to comply with scheduled visits, treatment plan, and follow up with research staff
* Age ≥ 21 years

Exclusion Criteria:

* Inability to comply taking NET
* Inability to comply to study procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Response to neoadjuvant endocrine therapy (NET) | From enrollment to the end of treatment at <=52 weeks
  Response to neoadjuvant endocrine therapy is defined as clear margins (defined as greater than 1mm) measured in the surgical pathology report. The proportion of women in each cohort with response will be estimated with exact 95% binomial confidence intervals.

SECONDARY OUTCOMES:
Physicians will predict PEPI score after NET for subjects enrolled in cohort B or C | From enrollment to the end of treatment at <=52 weeks
  * PEPI score is determined from surgical pathology report
  * Physicians can predict the PEPI score and drop in Ki-67 based on tumor size, biology, and patient preference for duration pre-NET. See chart:
  Surgical factors PEPI Score Tumor size T1/T2 1 T3/T3 3 Node Size Negative 0 Positive 3 Ki67 Level 0-2.7% 0 >2.7-7.3% 1 >7.3-19.7% 1 >19.7-53.1% 2 >53.1% 3 ER Status Negative 3
  • The physicians will be asked to predict whether the PEPI score post-surgery will be 0 (low risk of recurrence), 1 - 3 (intermediate risk of recurrence), > 4 (high risk of recurrence).
  The chart above is used clarify how physicians will at the subject's PEPI score.
Physicians will predict Ki67 after NET | From enrollment to the end of treatment at <=52 weeks
  * Ki67 is assessed by pathologist in the tumor specimen obtained from surgical resection
  * Physicians will be asked to predict whether Ki-67 post-surgery will fall below 15% (high proliferation fraction). (see chart above for breakdown of surgical factors and PEPI score).
  * Concordance between the physician prediction and post-surgery PEPI values will be assessed using the kappa statistic. Concordance will be assessed using the kappa statistic. Thirty women per cohort will allow estimation of the percent with response to NET with standard error < 0.10.

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington-Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided